CLINICAL TRIAL: NCT05875818
Title: Comparison of Effects of Tele-rehabilitation Versus In-clinic Rehabilitation for Upper Limb Motor Function in Chronic Stroke Patients
Brief Title: Comparison of Tele-rehabilitation Versus In-clinic Rehabilitation for Upper Limb Motor Function Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/542
Record Dates: First submitted 2023-03-18; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation (Other)
  Interventions: Diagnostic Test: Tele-rehabilitation
- In-clinic Rehabilitation (Experimental)
  Interventions: Diagnostic Test: In-clinic Rehabilitation

INTERVENTIONS:
Diagnostic Test: In-clinic Rehabilitation — Effects of In-clinic Rehabilitation for Upper Limb Motor Function in Chronic Stroke Patients
  Arms: In-clinic Rehabilitation
Diagnostic Test: Tele-rehabilitation — Effects of Tele-rehabilitation for Upper Limb Motor Function in Chronic Stroke Patients
  Arms: Tele-rehabilitation

SUMMARY:
To determine the effects of Tele-rehabilitation versus in-clinical rehabilitation for upper limb motor function and spasticity in chronic ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* • Patients from both genders.

  * Patients with chronic ischemic stroke i.e. 6 months or more.
  * Patients with 45 years old and above.
  * On modified Ashworth scale, patient with limb spasticity equal to 2 or less than 2.
  * On Mini Mental State Examination (MMSE), patients with good cognitive function minimum 24 or more.

Exclusion Criteria:

* • Patients with any recurrent stroke history.

  * Cognitive deficit patients (on Folstein Mini Mental state Examination score of less than 24)
  * Patient having other neurological diseases.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Fugal Myer assessment scale (FMAS) | 6 Months
  Fugal Myer assessment scale (FMAS) to check the pain and funcationality in stroke
Modified Ashworth Scale (MAS) | 6 Months
  Modified Ashworth Scale (MAS) to check the pain and funcationality in stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No